CLINICAL TRIAL: NCT00090688
Title: Safety and Immunogenicity of Oral Microencapsulated CS6 Vaccine and LT(R192G) Adjuvant in Volunteers
Brief Title: Phase 1 meCS6 + LT(R192G) Vaccine Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IND was terminated for being inactive for more than five years
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WRAIR 1065; HSRRB A-12367
Record Dates: First submitted 2004-09-02; First posted 2004-09-03 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2006-01

CONDITIONS: Diarrhea
Keywords: diarrhea
MeSH Terms: conditions — Diarrhea

INTERVENTIONS:
Biological: meCS6 + LT(R192G)

SUMMARY:
The study will enroll approximately 60 volunteers. The vaccine is given as a drink in flavored soda water. Volunteers will either receive a 3-dose vaccination with doses spaced two weeks apart or a 4-dose vaccination with doses spaced 2 days apart depending upon their availability for follow-up.

Once assigned to a vaccination schedule, volunteers will be randomly assigned to receive the meCS6 vaccine with or without the mLT adjuvant for all vaccine doses. Neither the study investigators nor the volunteers will know which group they are assigned.

Volunteers will be asked to be available for clinic visits and telephone follow-ups during the study period and provide blood and stool specimens for testing.

DETAILED DESCRIPTION:
The Phase 1 section of this study is a randomized double blind trial in which a total of 60 subjects (minimum of 52 allowable) will receive on of two oral vaccine doses according to the following chart:

Group Subset N CS6(Encapsulated) LT(R192G) I A 15 0.95mg 2 micrograms II B 15 0.95mg -- III A 15 0.95mg 2 micrograms IV B 15 0.95mg --

*minimum of 13 volunteers/group

Volunteers in Group I will receive three immunizations (study days 0, 14, and 28) during the vaccine series. Volunteers in Group II will receive four immunizations (study days 0, 2, 4, and 6) during the vaccine series. The two groups will be vaccinated separately for logistical purposes. Blood and stool specimens will be collected at intervals to examine systemic and mucosal vaccine antigen-specific immune responses. Vaccine safety will be actively evaluated during vaccination and for 4 weeks following the final vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* Available for required follow-up period
* Women must have a negative pregnancy test
* Women must not to try to become pregnant while on study and for 2 months after study is completed

Exclusion Criteria:

* History of travellers' diarrhea
* Occupation that involves handling of E. coli or cholera bacteria, or E. coli vaccine
* Regular use of anti-diarrheal, anti-constipation, or antacid therapy
* Abnormal bowel habits
* Pregnant or nursing women
* History of chronic gastrointestinal illness or major gastrointestinal surgery
* Allergies to vaccines
* Positive HIV, Hepatitis B or Hepatitis C tests
* Regular use of oral steroid medication
* Clinically significant abnormalities on physical examination

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2004-08

PRIMARY OUTCOMES:
Safety
Mucosal Immunogenicity
Systemic Immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Lapa, MD, Principal Investigator — Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States